CLINICAL TRIAL: NCT04069897
Title: Botulinum Toxin Type A Blockade of the Sphenopalatine Ganglion in Treatment-refractory Chronic Migraine
Acronym: MiBlock
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Oslo University Hospital (Other); Haukeland University Hospital (Other); Nordlandssykehuset HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/2161; 2018-004053-24 (EudraCT Number)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Migraine Disorders
Keywords: Botulinum Toxin Type A; Sphenopalatine Ganglion Block; Autonomic Nerve Block; Injections
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Idoxuridine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injections towards SPG (Experimental): Botulinum Toxin type A injections
  Interventions: Drug: Botulinum toxin type A
- Controls (Placebo Comparator): Placebo injections
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin 25 Allergan units in 0.5 ml Sodium Chloride (NaCl) 0.9 % Braun. Two injections, one in each side of the face, and targeting the sphenopalatine ganglion.
  Other Names: botox; Allergan
  Arms: Botox injections towards SPG
Drug: placebo — 0.5 ml Sodium Chloride (NaCl) 0.9% Braun. Two injections, one in each side of the face, and targeting the sphenopalatine ganglion.
  Other Names: sodium chloride
  Arms: Controls

SUMMARY:
This is a clinical trial to assess the efficacy of botox treatment of the sphenopalatine ganglion as an add-on treatment in drug resistant migraine. An injection targeting the ganglion is made possible by an image-guided device developed specifically for this purpose (MultiGuide) Study participants will be randomized to either placebo or botox after a 4 week run-in period. First, one injection will be given towards both the right and the left ganglion. After that there will be a follow-up of 12 weeks for efficacy and safety evaluation. The main efficacy measure is change in number of moderate to severe headache days before and after injection.

ELIGIBILITY:
Inclusion Criteria:

The participants must meet all of the inclusion criteria to participate in this study:

1. Informed and written consent.
2. Male or female, between 18 and 70 years of age
3. Masters a Scandinavian language at level sufficient to fully understand the written and verbal study information
4. Migraine, with or without aura, fulfilling the International Classification of Headache Disorders (ICHD) III criteria 1.3. for chronic migraine at time of inclusion
5. Chronic migraine at least for a period of 1 year prior to inclusion
6. Debut of episodic migraine before the age of 50, and chronic migraine before the age of 65.
7. The condition is pharmacologically refractory as defined in this study as insufficient treatment effect, contraindication(s) or intolerable side effect(s) of at least 3 medications from at least 2 of the following medication (drug) classes

   1. Beta-blockers
   2. RA(A)S-inhibitors
   3. Calcium-antagonists
   4. Antiepileptic drugs
   5. Tricyclic antidepressants
   6. Botulinum toxin A
   7. CGRP antagonists
8. Subject has had no change in type, dosage or dose frequency of preventive headache medications < 3 months prior to baseline/screening, or a minimum of 5 half-lives, whichever is longer.
9. Subject agrees to maintain current preventive headache medication regimens (no change in type, frequency, or dose) during the whole study period.
10. In the case of women of childbearing potential (WOCBP) they have to commit to highly effective contraception in a period of 4 weeks after injection (for details, confer section 4.3)
11. Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

All candidates meeting any of the exclusion criteria at baseline or visit 2 will be excluded from study participation:

1. Allergy or hypersensitivity reactions to marcaine, lidocaine, xylocaine, adrenaline, any botulinum toxin or similar substances.
2. Subject is unable to differentiate migraine from other concomitant headaches.
3. Subject with secondary headache conditions, with the exception of medication overuse headache.
4. Non-responder in regular clinical practice to preventive medications from ≥6 of the following 7 drug classes:

   1. Beta-blockers
   2. RA(A)S-inhibitors
   3. Calcium-antagonists
   4. Antiepileptic drugs
   5. Tricyclic antidepressants
   6. Botulinum toxin A
   7. CGRP antagonists
5. Subject has had a change in type, dosage or dose frequency of preventive headache medications < 3 months prior to baseline/screening, or a minimum of 5 half-lives, whichever is longer.
6. Subject has had a change in type, dosage or dose frequency of preventive headache medications during the baseline period, eg. prior to IMP administration
7. Botulinum toxin injections in the head and neck region, as part of migraine treatment or otherwise indicated on medical or cosmetic grounds, in the last 4 months before inclusion.
8. The discontinuation of CGRP-antagonists within 3 months before study inclusion or 5 half-lives, whichever is longer,
9. Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months before study inclusion or 5 half-lives, whichever is longer.
10. Subject is currently participating or has participated in the last 3 months in another clinical study in which the subject has, is, or will be exposed to an investigational or non-investigational drug or device.
11. Subject has had previous radiofrequency ablation, balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of the trigeminal ganglion or any branch of the trigeminal nerve.
12. Subject has had previous radiofrequency ablation (including non-lesional pulsed radiofrequency), balloon compression, gamma knife, or chemical denervation (e.g. glycerol treatments) of the SPG.
13. Subject has had blocks of short-acting anaesthetics of the SPG in the last 3 months.
14. Subject is or has been treated with occipital nerve stimulation or deep brain stimulation.
15. Ongoing abuse of drugs (including narcotics) or alcohol.
16. More than 4 days of opioid use per month (including codeine and tramadol), and any use of barbiturates
17. Treatment with pharmacological substances prior to SPG-injection that may interact with BTA (aminoglycosides, spectinomycin, neuromuscular blockers, both depolarizing agents (such as succinylcholine) or non-depolarizing (tubocurarine derivates), and anticholinesterases).
18. Inadequate contraceptive use. Women of childbearing potential (WOCBP) who do not use highly effective contraception (HEC) or use other medication that may interact and/or otherwise reduce the efficacy of the contraceptive agents in use.
19. Subject has undergone facial surgery in the area of the pterygopalatine fossa or zygomaticomaxillary at the planned injection site that, in the opinion of the Investigator, may lead to an inability to properly conduct the procedure.
20. Facial anomaly or trauma which renders the procedure difficult.
21. Subject currently has an active oral or dental abscess or a local infection at the site of injection based on present symptoms.
22. Subject has been diagnosed with any major infectious processes such as osteomyelitis, or primary or secondary malignancies involving the face that have been active or required treatment in the past 6 months.
23. Patients with comorbid psychiatric disorders with psychotic or other symptoms making compliance with the study protocol difficult, at the discretion of the investigator
24. Patients exhibiting a high degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator
25. Patients with disorders that severely inhibits lacrimation, at the discretion of the investigator
26. Patients with previous ischemic cardiovascular and cerebrovascular disorder with, in the opinion of the investigator, a moderate to high risk of new ischemic episodes.
27. Known infection or history of human immunodeficiency virus, tuberculosis, or chronic hepatitis B or C infection.
28. Subject has a history of bleeding disorders or coagulopathy, that, in the opinion of the Investigator, may lead to an inability to properly conduct the procedure.
29. Unable to stop antithrombotic medication e.g. platelet aggregation inhibitors and/or anticoagulation therapy, prior to procedure.
30. The patient cannot participate or successfully complete the study, in the opinion of their healthcare provider or the investigator, for any of the following reasons:

    * mentally or legally incapacitated or unable to give consent for any reason
    * in custody due to an administrative or a legal decision, under tutelage, or being admitted to a sanatorium or social institution
    * has any other condition, which, in the opinion of the investigator, makes the patient inappropriate for inclusion in the study
31. The patient is a study centre employee who is directly involved in the study or the relative of such an employee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean monthly headache days at weeks 5 - 8 post intervention | week 5 through week 8 in the post-injection period
  Change from baseline to week 5-8 post-intervention in frequency of moderate to severe headache days. Headache episodes that qualify is in the study defined as headache pain duration of ≥4 hours with a peak severity of moderate or severe intensity, or of any severity or duration if the subject takes and responds to rescue medication.

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events in the treatment | week 1 through week 12 in the post-injection period
  All adverse events and serious adverse events occurring in the 3 months follow up are registered in an electronic CRF. Frequency of AE and SAE are compared between the placebo group and the treatment group
Change from baseline in the mean monthly migraine days in the treatment | week 5 through week 8 in the post-injection period
  A migraine day is defined as one day with headache pain fulfilling the ICHD3-criteria for migraine or probable migraine. However, a headache duration of less than 4 hours is allowed if the subject takes and responds to triptans. The frequency of headache days in the baseline period are compared to the frequency in week 5-8 post-intervention
number of treatment responders (≥ 30% reduction in mean monthly headache days) | week 5 through week 8 in the post-injection period
  A 30% treatment response is defined as a patient with a ≥ 30% reduction in frequency of headache days during weeks 5 - 8 post-intervention compared to baseline. Headache is defined as in the primary outcome, i.e. moderate to severe headache days. The number of responders is compared between the intervention and the placebo group
Change from baseline in the mean monthly headache intensity in the treatment | week 1 through week 4, week 5 through week 8 and week 9 through week 12 in the post-injection period
  Attack intensity is reported daily on a 11-point numerical response scale (NRS) in the electronic headache diary. The mean attack intensity in week 5 - 8 post-intervention is compared to baseline in the active group versus the placebo group.
Change from baseline in the mean monthly occurrence of cumulative hours per 28 days of moderate/severe pain in the treatment | : week 1 through week 4, week 5 through week 8 and week 9 through week 12 in the post-injection period
  The difference in hours with NRS ≥4 in the baseline period and weeks 1-4, 5-8 and 9-12 post injection are compared between the active group and the placebo group
Change from baseline in the mean monthly number of days with rescue medication in the treatment | : week 1 through week 4, week 5 through week 8 and week 9 through week 12 in the post-injection period
  Any use of rescue medication is reported in the headache diary every day. The number of days with registered use of any headache related rescue medication in weeks 1-4, 5-8 and 9-12 post-intervention is compared to the baseline period
Migraine specific quality of life questionnaire | week 8 and week 12 post-injection
  Study participants will fill in the 6-question Headache impact test (HIT-6) at visit 1 (at inclusion) and at week 8 and week 12 postintervention. Scores are compared between the placebo and the treatment group
Migraine specific quality of life questionnaire | week 8 and week 12 post-injection
  Study participants will fill in the 14-question Migraine-Specific Quality-of-Life Questionnaire Version 2.1 (MSQ) at visit 1 (at inclusion) and at week 8 and week 12 postintervention. Scores are compared between the placebo and the treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Geir Bråthen, md phd, Study Director — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, department of Neurology, Bergen
  - Nordland Hospital, department of Neurology, Bodø
  - Nevroklinikken Universitetet i Oslo, Oslo Universitetssykehus HF, Oslo
  - St Olavs Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared within 6 months after study results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 6 months after study results publication
Access Criteria: erling.tronvik@ntnu.no